CLINICAL TRIAL: NCT01198964
Title: U.S.-German Collaboration: Optimization of Human Cortical Stimulation
Brief Title: Optimization of Human Cortical Stimulation
Acronym: BCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jeffrey Ojemann, Professor, Neurological Surgery, University of Washington
Other Study IDs: STUDY00001800
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Epilepsy; Brain Injury
Keywords: ECoG; Epilepsy; cortical; stimulation; Electrocorticography; electrodes; mapping
MeSH Terms: conditions — Epilepsy; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epileptic Patients: The population of patients with medically refractory epilepsy will already have been recommended clinically for electrode grid placement on the brain and high-level stimulation to map brain function.
  Interventions: Procedure: Low-level cortical stimulation

INTERVENTIONS:
Procedure: Low-level cortical stimulation — A couple of electrodes will be stimulated (at a lower level than the stimulation used for standard care) over a period of 4-12 hours based on the signals defined by the motor or language task.

SUMMARY:
We will observe epileptic patients who already have electrodes implanted on the brain and are receiving high-level brain stimulation for clinical purposes while testing their motor and language function. We propose to do a limited, low-level brain stimulation to show that the signatures of local activity in the target area change as an effect of brain stimulation. The goal of this study is to understand the feasibility of a novel recurrent brain-computer interface that could eventually promote targeted functional recovery in subjects who have had a brain injury.

DETAILED DESCRIPTION:
The subject will have already been scheduled for placement of the ECoG electrodes on the surface of the brain and who will, for all clinical purposes, subsequently receive stimulation for mapping of function of the ECoG sites. The decision to place the electrodes on the brain, the location of the electrodes and the length of time the electrodes are in are all part of clinical care.

There will be two types of testing, motor and language. Motor will involve inducing stimulation to the thumb cortex and the wrist cortex. There will be a conditioning of this over 4-12 hours. Language will involve showing pictures on a computer screen and the subject will be observed whether speech is disrupted with stimulation or not.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Male and Female
* Able to understand English for consenting and testing
* Referred for surgical implantation of electrodes

Exclusion Criteria:

* Under 18 years of age
* Pregnant women
* Prisoners
* Mentally disabled IQ < 70
* Non English Speaking
* Not candidates for surgical implantation of electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 18 and older male and female epileptic patients who are referred for surgical implantation of electrodes.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2010-09; Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Link EMG activity produced during a motor task to stimulation of a part of the brain | 5 years
  Attempt to link EMG activity produced during a motor task to stimulation of a part of the brain nearby, but distinct from, the part of the brain normally used to perform the task.

SECONDARY OUTCOMES:
Evaluate distribution of current from stimulation | 5 years
  Using mathematical models to determine if current is going to areas expected

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G Ojemann, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- See also: Home page for Harborview's Regional Epilepsy Center — http://pcs.hmc.washington.edu/epilepsy/